CLINICAL TRIAL: NCT03767556
Title: Effects of Respiratory Muscle Training on Lung Function, Respiratory Muscle Function and Physical Fitness in Obese Women
Brief Title: Effects of Respiratory Muscle Training in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Eli Maria Pazzianotto Forti, Principal Investigador, Universidade Metodista de Piracicaba
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Tamires2018
Record Dates: First submitted 2018-10-17; First posted 2018-12-06 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Inadequate or Impaired Respiratory Function; Diabetes; Hypertension
Keywords: physical tests; functional capacity; spirometry; travelled distance; cardiorespiratory fitness; flexibility; respiratory pressures; dyspnea
MeSH Terms: conditions — Respiratory Insufficiency; Diabetes Mellitus; Hypertension; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will not receive intervention
- Inspiratory Muscle Training (Experimental): This group, for inspiratory muscle training, will use the Powerbreathe® K5 device. This device will be adjusted with a load of 55% of previously assessed MIP. The volunteer will be instructed to inhale with sufficient force to overcome the resistance of the equipment and subsequently perform a normal expiration. During the 4-week period of respiratory muscle training volunteers will be instructed to perform 2 sets with 30 inspiratory efforts, 5 days a week. The training load will be readjusted on the first day of training each week, after a new reassessment of the PIMax in order to guarantee the overload during inspiratory muscle training.
  Interventions: Procedure: Inspiratory muscle training

INTERVENTIONS:
Procedure: Inspiratory muscle training — Powerbreathe® K5
  Arms: Inspiratory Muscle Training

SUMMARY:
The objective of this study will be to evaluate the effects of inspiratory muscle training (IMT) on the physical fitness of obese women

It is believed that the application of these exercises helps in the improvement of inspiratory muscle performance, which should improve physical fitness and thus allow a better performance in the activities of daily living.

DETAILED DESCRIPTION:
This is a clinical trial, in which adult obese volunteers aged 20-59 years will be evaluated, which will be randomized into two groups: training group (GT) and control group (CG). Both groups should meet the following inclusion criteria: Age between 20 and 59 years, BMI> 35 and <55 kg / m², with clinical stability, able to perform the physical tests and acceptance to participate in the study. Women with reports of decompensated heart disease, chronic obstructive pulmonary disease and asthma will be excluded; musculoskeletal and / or neuromuscular changes, which make it impossible to perform the tests. The evaluations will occur in two days with at least 48 hours of interval between them, within a period of seven days, before and after the respiratory muscle training of four weeks. In addition to anamnesis, the initial evaluation will include assessment of pulmonary function (SLF, forced vital capacity (FVC) and maximal voluntary ventilation (VVM)) by spirometry; respiratory muscle evaluation through the measures of Maximum Inspiratory Pressure (PIMax) and maximal sustained inspiratory pressure (PIMaxS); physical fitness assessment through the 6-minute step test (TD6), incremental shuttle walking test (ISWT) and Sentar e Levantar (SL) test, as well as assessment of dyspnea. For the TMI will be used equipment with pressure threshold pressure. During the 4-week period, the IMT will be performed 5 days a week and will consist of 2 series with 30 inspirations. Inspirations will be performed slowly and protracted. The training load will be 55% of the PIMáx readjusted weekly. Statistical analysis will be performed using BioEstat version 5.3. To evaluate the normality of distribution of the data will be used Shapiro-Wilk test. For the comparison of all variables studied, the Student's t-test or the Mann-Wittney test will be used. Pre- and post-training parametric results will also be compared statistically using variance analyzes of two variables (group × time) (ANOVA). Bonferroni tests will be used to examine differences between groups when indicated by ANOVA. The significance level of 5% will be adopted for all analyzes (P <0.05) where the data will be expressed as mean and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* BMI> 35 and <55 kg / m²
* with clinical stability
* suitable for physical tests
* acceptance to participate in the study

Exclusion Criteria:

* women with reports of decompensated heart disease
* chronic obstructive pulmonary disease and asthma
* musculoskeletal and / or neuromuscular changes,
* which make it impossible to perform the tests.

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
EVALUATION OF LUNG VOLUMES AND CAPACITIES | before and after the intervention, for 2 days with a 72-hour interval
  Spirometry will be out according to the guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS) (2005). The values extracted will be selected according to Pereira (2002), and the predicted values calculated using the equation proposed by Pereira et al. (1992) for Brazilians.

SECONDARY OUTCOMES:
EVALUATION OF PHYSICAL ACTIVITY LEVEL | before and after the intervention, for 2 days with a 72-hour interval
  Volunteers will respond to the International Physical Activity Questionnaire, which is an instrument that allows estimating the weekly time spent in physical activity. The final classification given by the International Physical Activity Questionnaire occurs in five levels of physical activity: Very Active, Active, Irregularly active and Sedentary.
6-MINUTE DEGREE TEST (TD6) | before and after the intervention, for 2 days with a 72-hour interval
  The TD6 will be used for the evaluation of cardiorespiratory fitness by calculating the maximum oxygen consumption (VO2 max) in an indirect way and the functional capacity of the volunteers. The TD6 outcome will be the number of volunteer climbs on the rung (PESSOA et al., 2015). The values reached in the number and the rhythm of ascents in the step will express the functional capacity.
INCREMENTAL SHUTTLE WALKING TEST (ISWT) | before and after the intervention, for 2 days with a 72-hour interval
  The ISWT will be used to determine the functional capacity of the volunteers by the distance traveled during the test. It is a walking test, with progressive loading, given by the increase in walking speed required to overcome each stage of the test. The ISWT will be controlled by specific software, which determines the speed and pace of each stage of the test. This test will be carried out in a corridor in which 10 meters in length, delimited by cones, at each end, will be demarcated by volunteers, obeying each sound signal programmed by Sing et al. (1992). The test will be terminated at the signal of inability to continue or non-accompaniment of speeds by the volunteer.
TEST TO SIT AND LIFT | before and after the intervention, for 2 days with a 72-hour interval
  This test will be used to determine the indirect force in the lower limbs. To perform this test, a chair with a height of 40 cm will be used, with backrest, in which the volunteer will begin the test in the sitting position, in the middle of the seat, with the spine erect, feet resting on the floor and the arms crossed against the thorax. At the investigator's signal, the volunteer should stand up, stand fully up, and then return to the seated position. Volunteers will be encouraged to sit and stand up as often as possible in 30 seconds. The result will be determined by counting the number of times the volunteer correctly performed the movements of sitting and lifting of the chair without the aid of the movement of the upper limbs
EVALUATION OF INSPIRATORY MUSCLE STRENGTH | before and after the intervention, for 2 days with a 72-hour interval
  The Maximum Inspiratory Pressure (PIMax) and Maximum Expiratory Pressure (PEMax) measurements will be performed. The measures of the MIP will aim beyond the evaluation of the strength of the respiratory muscles, establish the initial load of the resistance test of the respiratory muscles as well as the training load. The measurements of PImax and PEmax, will be evaluated through an analog manovacuometer. Each participant should perform three to five maximum inspiratory and reproducible inspiratory efforts provided there has been a maximum difference of 10% between them being the highest value considered for statistical analysis. The time interval between consecutive measurements was 1 minute.

CONTACTS AND LOCATIONS:
Overall Officials: Eli M Pazzianoto-Forti, Phd, Principal Investigator — Universidade Metodista de Piracicaba
Locations (1):
- Universidade Metodista de Piracicaba (UNIMEP), Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No